CLINICAL TRIAL: NCT05508828
Title: Early Percutaneous Continuous Irrigation Assisted Vacuum Drainage Combined With Transgastric Necrosectomy Using Lumen Apposing Metal Stents in Treatment of Severe Acute Pancreatitis
Brief Title: Percutaneous Continuous Irrigation Combined With Transgastric Necrosectomy usingLAMS in Treatment of SAP
Acronym: PCISLAMS
Status: Completed | Type: Observational
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Other Study IDs: DRUMPCILAMS
Record Dates: First submitted 2022-08-14; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2019-01

CONDITIONS: Severe Acute Pancreatitis; Pancreatic Necrosis
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study group: We retrospectively analysis of 8 consecutive patients with SAP and IPN. SAP was diagnosed with persistent organ failure >48h. IPN was considered when the following situations occur: ≥38.5℃; increasing WBC, CRP or procalcitonin; rapid clinical deterioration; signs of gas was present in areas of necrosis.
  Interventions: Procedure: Percutaneous Continuous Irrigation assisted Vacuum Drainage Combined With Transgastric Necrosectomy

INTERVENTIONS:
Procedure: Percutaneous Continuous Irrigation assisted Vacuum Drainage Combined With Transgastric Necrosectomy — All patients with SAP were given contrast enhanced CT scan within 48 hours after admission to identify the location and range of the necrosis. If the patient's condition progressively worsened, a multifunctional irrigation-assisted vacuum drainage tube was placed by the CT-guided Seldinger technique in each of the necrosis cavity. Subsequently, transgastric necrosectomy were performed by one or two experienced endoscopist under conscious sedation. The procedure was repeated until all loosely adherent necrotic material were cleared and replaced by granulation tissue. Percutaneous irrigation was stopped and replace with simple drainage if the patient's condition continues to improved and the cavity confirmed by CT was resolution. If the drainage volume was less than 10 mL/day for 3 consecutive days, clamp the drainage tube and remove it finally.

SUMMARY:
Severe acute pancreatitis (SAP) is the most severe form of acute pancreatitis (AP) and Infection of pancreatic necrosis (IPN) have shown to be one of the decisive factors defining the severity of illness.

Minimally invasive techniques including endoscopy, laparoscopy, retroperitoneal approaches, etc., have recently been widely used for debridement because the procedure can further reduces surgical stress and performed not require general anesthesia, thereby reducing complications. Studies have shown that endoscopic transgastric necrosectomy can significantly reduced the proinflammatory response, complications, and hospital stay. Despite these advantages, there are some limitations with this approach. First, transgastric necrosectomy should be performed as late (about 4 weeks) in the course of the disease as possible to allow necrosis to wrap, since early debridement may result in a higher patient fatality rate. However, patients with SAP are often in a severely ill state due to sepsis or MODS at an early stage, which causes them unable to adhere to necrotic tissue encapsulation by conservative treatment. Second, the ideal patient to select for this approach has necrosis confined in the vicinity of gastroduodenal location. Last, up to 27% of IPN patients require additional percutaneous catheter drainage (PCD) after undergoing endoscopic transluminal therapy. This may be explained by the fact that dissemination of necrosis, digestive enzymes and inflammatory mediators from the necrotic tissue lumen to other parts of the abdominal cavity during endoscopic procedures.

Percutaneous catheter drainage (PCD) has always been the principal treatment measure for patients with AP at early stage (< 4 weeks) or those with collections or necrosis extending into deeper anatomical planes. Irrigation through peripancreatic drainage placed after open laparotomy has been the standard treatment for patients with AP who had undergone surgical necrosectomy. However, this proactive approach has not been widely used in the setting of PCD.

To adequate drainage and removal of necrosis, an early percutaneous continuous irrigation assisted vacuum drainage in combination with subsequent endoscopic transgastric necrosectomy which has not been reported so far was applied in critically ill patients with SAP.

DETAILED DESCRIPTION:
Severe Acute Pancreatitis (SAP) Treatment Protocol After admission, patients were given intravenous analgetics, omeprazole and somatostatin, and nasojejunal tubes were placed for EN. Once fever developed, broad-spectrum antibiotics were given empirically. If the patient was concomitant with shock, respiratory failure, and acute kidney injury, appropriate organ support was provided. Patients with biliary pancreatitis was given encoscopic retrograde cholangiopancreato graphy (ERCP) within 24 h after admission. When the patient was diagnosed with hyperlipidemic pancreatitis and plasma triglyceride ≥11.3 mmol/L, plasma exchange was administered immediately. All patients were given contrast enhanced CT within 48 hours after admission to identify the location and range of the necrosis and calculate the CT severity index (CISI).

Procedure All PCD and endoscopic procedures were performed under conscious sedation or local anesthesia. If the patient's condition progressively worsened, a multifunctional irrigation-assisted vacuum drainage tube was placed by the CT-guided Seldinger technique in each of the necrosis cavity. The tube was administered with continuous internal irrigation and vacuum drainage as described in below: (1) the end of the drainage tube (the adapter) was connected to a vacuum device that delivers a controlled negative pressure within the range of 8-10 kPa. (2) a large volume of 0.9% normal saline was infused into the necrosis cavity constantly (1500mL a day, 65mL an hour) through the durg entrance, allowing for continuous irrigation; (3) the inside drainage tube was flush by rapid manual injection of 50-100 mL 0.9% normal saline twice a day through the drug entrance and inject 20-50 mL of 0.9% normal saline daily through water entrance to prevent the tube from becoming blocked by necrosis, debris or omentum; (4) total irrigation and drainage volume were checked every 8 hours to keep the irrigation-drainage balanced. All tubes were checked daily and replaced when the tube was translocated or blocked. When the volume of irrigation exceeds the drainage 500 mL/day or if there were serious complications associated with the drainage tube, continuous irrigation and vacuum drainage should be stopped immediately and the tube was the traditional drainage was performed.

Approximately 4 weeks after disease onset or the formation of well-defined wall was confirmed by repeat CT scan, transgastric necrosectomy were performed by one or two experienced endoscopist under conscious sedation. Transgastric necrosectomy was repeated, mostly every three to five days, until all loosely adherent necrotic material were cleared and replaced by granulation tissue. In the course of the procedure, antibiotic administration was adjusted based on the results of the microbiological culture results. Subsequently, percutaneous irrigation was stopped and replace with simple drainage if the patient's condition continues to improved and the cavity confirmed by CT was resolution. If the drainage volume was less than 10 mL/day for 3 consecutive days, clamp the drainage tube and remove it finally.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with SAP
* Concurrent IPN

Exclusion Criteria:

* Age <18 years or > 80 years
* Patients or family members disagreed with this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with SAP and IPN;SAP was diagnosed according to the revised Atlanta classification, which defined simultaneous persistent single or multiple organ failure >48h;IPN was considered when the following situations occur: persistent fever ≥38.5℃; increasing blood white blood cells (WBC), C-reactive protein (CRP) or procalcitonin; rapid deterioration of clinical deterioration; signs of gas was present in areas of necrosis. IPN is confirmed when the patient undergoes fine needle aspiration and the culture was positive.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-08-14 (Actual)

PRIMARY OUTCOMES:
mortality | Day28 after enrollment
  28day-mortality

SECONDARY OUTCOMES:
PCD | From the first catheter placement to total catheter removal
  duration of PCD
endoscopic procedures | through study completion, an average of 3 months
  number of endoscopic procedures

CONTACTS AND LOCATIONS:
Overall Officials: Wenkui Yu, Ph.D, Study Chair — Study concept and study design
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van Santvoort HC, Besselink MG, Bakker OJ, Hofker HS, Boermeester MA, Dejong CH, van Goor H, Schaapherder AF, van Eijck CH, Bollen TL, van Ramshorst B, Nieuwenhuijs VB, Timmer R, Lameris JS, Kruyt PM, Manusama ER, van der Harst E, van der Schelling GP, Karsten T, Hesselink EJ, van Laarhoven CJ, Rosman C, Bosscha K, de Wit RJ, Houdijk AP, van Leeuwen MS, Buskens E, Gooszen HG; Dutch Pancreatitis Study Group. A step-up approach or open necrosectomy for necrotizing pancreatitis. N Engl J Med. 2010 Apr 22;362(16):1491-502. doi: 10.1056/NEJMoa0908821. PMID 20410514
- [Result] Lee JK, Kwak KK, Park JK, Yoon WJ, Lee SH, Ryu JK, Kim YT, Yoon YB. The efficacy of nonsurgical treatment of infected pancreatic necrosis. Pancreas. 2007 May;34(4):399-404. doi: 10.1097/MPA.0b013e318043c0b1. PMID 17446837
- [Result] Ross A, Gluck M, Irani S, Hauptmann E, Fotoohi M, Siegal J, Robinson D, Crane R, Kozarek R. Combined endoscopic and percutaneous drainage of organized pancreatic necrosis. Gastrointest Endosc. 2010 Jan;71(1):79-84. doi: 10.1016/j.gie.2009.06.037. Epub 2009 Oct 27. PMID 19863956
- [Result] Sahar N, Kozarek R, Kanji ZS, Ross AS, Gluck M, Gan SI, Larsen M, Irani S. Do lumen-apposing metal stents (LAMS) improve treatment outcomes of walled-off pancreatic necrosis over plastic stents using dual-modality drainage? Endosc Int Open. 2017 Nov;5(11):E1052-E1059. doi: 10.1055/s-0043-111794. Epub 2017 Oct 26. PMID 29090245
- [Result] Jagielski M, Smoczynski M, Studniarek M, Adrych K. Endoscopic drainage combined with percutaneous drainage in treatment of walled-off pancreatic necrosis - a single-center experience. Prz Gastroenterol. 2018;13(2):137-142. doi: 10.5114/pg.2018.72604. Epub 2018 Jan 5. PMID 30002773
- [Derived] Zhang B, Gao T, Wang Y, Zhu H, Liu S, Chen M, Yu W, Zhu Z. A novel mini-invasive step-up approach for the treatment of severe acute pancreatitis with extensive infected necrosis: A single center case series study. Medicine (Baltimore). 2023 Mar 17;102(11):e33288. doi: 10.1097/MD.0000000000033288. PMID 36930105